CLINICAL TRIAL: NCT05524311
Title: Baricitinib in the Treatment of New-onset Juvenile Dermatomyositis
Brief Title: Baricitinib in the Treatment of New-onset Juvenile Dermatomyositis (MYOCIT)
Acronym: MYOCIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP211036; 2022-000506-10 (EudraCT Number)
Record Dates: First submitted 2022-07-05; First posted 2022-09-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Juvenile Dermatomyositis
Keywords: juvenile dermatomyositis; baricitinib
MeSH Terms: conditions — Dermatomyositis | interventions — baricitinib; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental)
  Interventions: Drug: Baricitinib; Biological: pharmacokinetics study; Biological: dosage of cytokines; Biological: transcriptomic analysis; Behavioral: Parent version of the Child Health Questionnaire (CHQ); Behavioral: Childhood Health Assessment Questionnaire; Biological: Pregnancy test

INTERVENTIONS:
Drug: Baricitinib — Oral tablets (2 mg) will be used For children > or = 6 years: 4 mg once a day (2 x 2 mg) during the 24 weeks-period study For children < 6 years: 2 mg once a day during the 24 weeks -period study
Biological: pharmacokinetics study — additionnal blood sampling at week 4, 8, 12, and 24
Biological: dosage of cytokines — additionnal blood sampling at weeks 0, 4 and 24
Biological: transcriptomic analysis — additionnal blood sampling at weeks 0, 4 and 24
Behavioral: Parent version of the Child Health Questionnaire (CHQ) — Evaluate by parents at each visits
Behavioral: Childhood Health Assessment Questionnaire — Evaluate by parents at each visits
Biological: Pregnancy test — Urine pregnancy test at V4 A dosage of bHCG with current biological analysis is done at each visit (except V4)

SUMMARY:
The MYOCIT study aims to evaluate the efficacy and safety of baricitinib in association with corticosteroids in new-onset patients with juvenile dermatomyositis (JDM) in a phase II trial with the objective to obtain a better efficacy than the conventional combination methotrexate (MTX) and corticosteroids over the 24 week study period. Thus, the investigators hypothesize that baricitinib could be used as a first line treatment in all forms of DMJ, including the most severe one, with a good safety profile.

DETAILED DESCRIPTION:
Juvenile dermatomyositis (JDM) is a rare and severe paediatric-onset idiopathic inflammatory myopathy, associated with significant morbidity and mortality. The combination of corticosteroids and methotrexate (MTX) is recommended in new-onset JDM according to one randomized trial. However, in this trial, treatment failures were reported in 13/46 (28%) patients and severe JDM, (cutaneous or gastrointestinal ulceration, interstitial pulmonary disease, cardiomyopathy) were not taken into account. These data emphasize the need for a more efficient first-line treatment. Considering: 1) the strong implication of type IFN-I in the pathophysiology of JDM 2) the report of the efficacy and safety of JAK inhibitors (JAKis) (baricitinb, tofacitinib) in about 50 refractory DM patients, and 9 JDM, a trial which evaluates the efficacy and safety of baricitinib in combination with corticosteroids in new-onset JDM is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 3-18 years with new-onset juvenile dermatomyositis, according to the ENMC 2018 dermatomyositis classification criteria
* Muscle weakness at MMT and/or CMAS (MMT < 74 and/or CMAS < 45)
* Seropositivity or vaccination for chickenpox
* For patients of childbearing age (following menarche) : Negative βHCG and effective method of contraception (sexual abstinence, hormonal contraception, intrauterine device or hormone-releasing system, cap, diaphragm or sponge with spermicide, condom) until the 7 days after administration of the last dose of Baricitinib
* Informed consent form signed by the patient or child' s parents Patient affiliated to a social security regime

Exclusion Criteria

* Amyopathic dermatomyositis (without muscle weakness)
* Inability to be treated by oral way or to take pills
* Previous treatment with JAK inhibitor
* Previous treatment of JDM with immunosuppressive drugs or biologics other than corticosteroids. Previous treatment with prednisone was allowed for no more than 1 month.
* Previous history of cancer
* Live vaccine within the 4 weeks before starting baricitinib therapy
* Current, or recent (< 4 weeks prior to baseline) of active infections according to investigator appreciation, but necessarily, including HBV, HCV, HIV, tuberculosis.
* Positive blood CMV PCR
* Creatinine clearance < 40 ml/min
* Lymphocytes < 0,5x109 cell/L and Neutrophils < 1x109 cell/L
* Hemoglobin < 8 g/dL
* Symptomatic herpes herpes simplex infection within 12 weeks prior to inclusion
* History of thrombosis or considered at high risk of venous thrombosis by the investigator
* Presence of severe JDM-related involvements: cardiovascular (requiring vasopressive drug and/or intensive care unit), respiratory (requiring oxygen and/or intensive care unit), gastrointestinal (requiring abdominal surgery).
* History of severe non-related JDM involvement: cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological or neuropsychiatric disorders or any other serious and/or instable illness that, in the opinion of the investigator, could constitute an unacceptable risk, when taking baricitinib.
* Actual or in project of pregrancy and breast-feeding until the 7 days after administration of the last dose of Baricitinib
* Patient on AME (state medical aid)
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
PRINTO 20 (Paediatric Rheumatology INternational Trials Organisation scale) | At week 24
  Achievement of the validated juvenile dermatomyositis PRINTO 20 level of improvement. PRINTO 20 level of improvement is defined as a 20% or greater improvement in three or more of the six variables of the juvenile dermatomyositis core set, with one or no variable worsening by more than 30% (muscle strength can not be the variable worsening) :
  1. muscle strength, assessed with the Childhood Myositis Assessment Scale (CMAS),
  2. physician's global assessment of the patient's disease activity (Physician's VAS)
  3. global disease activity assessment through the Disease Activity Score (DAS)
  4. functional ability through the Childhood Health Assessment Questionnaire (C-HAQ)
  5. parent's global assessment of the child's overall wellbeing (Parent's VAS)
  6. health-related quality of life, through the parent version of the Child Health Questionnaire (CHQ-Phs) A higher score is 100% and means a better outcome, a lower score is 0% and means a worse result.

SECONDARY OUTCOMES:
PRINTO 20 Paediatric Rheumatology INternational Trials Organisation scale - level 20 | At week 4, 8, 12 and 16
  achievement of the validated juvenile dermatomyositis PRINTO 20 level ; reaching a minimum of 20 % a higher score is 100% and mean a better outcome a lower score is 0% and means a worse result
PRINTO 50 Paediatric Rheumatology INternational Trials Organisation scale - level 50 | At week 4, 8, 12 and 16
  achievement of the validated juvenile dermatomyositis PRINTO 50 level ; reaching a minimum of 50 % a higher score is 100% and mean a better outcome a lower score is 0% and means a worse result
PRINTO 70 Paediatric Rheumatology INternational Trials Organisation scale - level 70 | At week 4, 8, 12 and 16
  achievement of the validated juvenile dermatomyositis PRINTO 70 level ; reaching a minimum of 70 % a higher score is 100% and mean a better outcome a lower score is 0% and means a worse result
PRINTO 90 Paediatric Rheumatology INternational Trials Organisation scale - level 90 | At week 4, 8, 12 and 16
  achievement of the validated juvenile dermatomyositis PRINTO 90 level ; reaching a minimum of 90 % a higher score is 100% and mean a better outcome a lower score is 0% and means a worse result
Total Improvement Score (TIS) | At inclusion, weeks 4, 8, 12, 16 and 24
  Relative and absolute variations of TIS. The TIS is the sum of the improvement in each of the six core set measures of disease activits The minimum score is 0 (worse) and maximum score is 100 (better) A major response is defined by a score > 70 A moderate response is defined by a score > 45 A minimal response is defined by a score > 30
Clinically inactive disease | At weeks 4, 8, 12 and 24
  according to the PRINTO criteria
Cutaneous Dermatomyositis Disease Area and Severity Index (CDSAI) | At inclusion, weeks 4, 8, 12, 16 and 24
  assess skin activity and damage across multiple body regions in patients with dermatomyositis
Myositis Disease Activity Assessment VAS (MYOACT) | At inclusion, weeks 4, 8, 12, 16 and 24
  Assess Relative and absolute variations of extramuscular activity
interstitial lung disease | At inclusion and at week 24
  Assessed by improvement of at least 10% of FCV, PTC, and DLCO and/or improvement of Lung tomodensitomery according to a specific scale
Dose of corticosteroid | At week 24
  Dose tapering at 6 months
Pharmacokinetics study | At weeks 4, 8, 12, and 24
  Non-compartmental analysis of baricitinib
Pharmacokinetics (PK) study with area under the curve | At weeks 4, 8, 12, and 24
  Correlation between area under the curve AUC in ng.h/ml (PK parameter of baricitinib) and disease activity 's scores
Pharmacokinetics (PK) study with maximal concentration | At weeks 4, 8, 12, and 24
  Correlation between maximal concentration Cmax in ng/mL (PK parameter of baricitinib) and disease activity 's scores
Pharmacokinetics (PK) study with through concentration | At weeks 4, 8, 12, and 24
  Correlation between through concentration Ctrough, in ng/mL (PK parameter of baricitinib) and disease activity 's scores
dosage of cytokines | At inclusion, weeks 4 and 24
  Measurement of serum IFN -, IFN-γ, IL-1β, IL-4, Il-5, IL-6, IL-8, IL-10, IL-12p70, IL-22, TNF α
transcriptomic analysis | At inclusion, weeks 4 and 24
  Study of genes expression within 800 genes related to immunity
Biopsy | At inclusion, weeks 4 and 24
  Assessment of muscle biopsies according to the internationally validated score system

CONTACTS AND LOCATIONS:
Overall Officials: Cyril GITIAUX, Doctor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (13):
- France (13):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital La Timone, Marseille
  - Hôpital Villeneuce, Montpellier
  - Hôpital Brabois, Nancy
  - Hopital Necker - Enfants malades : unité d'immuno-hématologie et rhumatologie, Paris
  - Hôpital du Kremlin-Bicêtre, Paris
  - Hôpital Necker - Enfants malades : service de dermatologie, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Trousseau, Paris
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Purpan, Toulouse

REFERENCES:
- [Background] Ruperto N, Ravelli A, Pistorio A, Ferriani V, Calvo I, Ganser G, Brunner J, Dannecker G, Silva CA, Stanevicha V, Cate RT, van Suijlekom-Smit LW, Voygioyka O, Fischbach M, Foeldvari I, Hilario O, Modesto C, Saurenmann RK, Sauvain MJ, Scheibel I, Sommelet D, Tambic-Bukovac L, Barcellona R, Brik R, Ehl S, Jovanovic M, Rovensky J, Bagnasco F, Lovell DJ, Martini A; Paediatric Rheumatology International Trials Organisation (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). The provisional Paediatric Rheumatology International Trials Organisation/American College of Rheumatology/European League Against Rheumatism Disease activity core set for the evaluation of response to therapy in juvenile dermatomyositis: a prospective validation study. Arthritis Rheum. 2008 Jan 15;59(1):4-13. doi: 10.1002/art.23248. PMID 18163404
- [Background] Lazarevic D, Pistorio A, Palmisani E, Miettunen P, Ravelli A, Pilkington C, Wulffraat NM, Malattia C, Garay SM, Hofer M, Quartier P, Dolezalova P, Penades IC, Ferriani VP, Ganser G, Kasapcopur O, Melo-Gomes JA, Reed AM, Wierzbowska M, Rider LG, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). The PRINTO criteria for clinically inactive disease in juvenile dermatomyositis. Ann Rheum Dis. 2013 May;72(5):686-93. doi: 10.1136/annrheumdis-2012-201483. Epub 2012 Jun 26. PMID 22736096
- [Background] Bode RK, Klein-Gitelman MS, Miller ML, Lechman TS, Pachman LM. Disease activity score for children with juvenile dermatomyositis: reliability and validity evidence. Arthritis Rheum. 2003 Feb 15;49(1):7-15. doi: 10.1002/art.10924. PMID 12579588
- [Background] Giancane G, Lavarello C, Pistorio A, Oliveira SK, Zulian F, Cuttica R, Fischbach M, Magnusson B, Pastore S, Marini R, Martino S, Pagnier A, Soler C, Stanevicha V, Ten Cate R, Uziel Y, Vojinovic J, Fueri E, Ravelli A, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). The PRINTO evidence-based proposal for glucocorticoids tapering/discontinuation in new onset juvenile dermatomyositis patients. Pediatr Rheumatol Online J. 2019 May 22;17(1):24. doi: 10.1186/s12969-019-0326-5. PMID 31118099
- [Background] Mammen AL, Allenbach Y, Stenzel W, Benveniste O; ENMC 239th Workshop Study Group. 239th ENMC International Workshop: Classification of dermatomyositis, Amsterdam, the Netherlands, 14-16 December 2018. Neuromuscul Disord. 2020 Jan;30(1):70-92. doi: 10.1016/j.nmd.2019.10.005. Epub 2019 Oct 25. No abstract available. PMID 31791867
- [Background] Singh G, Athreya BH, Fries JF, Goldsmith DP. Measurement of health status in children with juvenile rheumatoid arthritis. Arthritis Rheum. 1994 Dec;37(12):1761-9. doi: 10.1002/art.1780371209. PMID 7986222